CLINICAL TRIAL: NCT04580797
Title: A PHASE 1, OPEN-LABEL STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE PHARMACOKINETICS OF PF-06700841 FOLLOWING SINGLE ORAL ADMINISTRATION OF MODIFIED RELEASE FORMULATIONS UNDER FED AND FASTED CONDITIONS IN PART A AND A RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO CONTROLLED STUDY TO EVALUATE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF PF-06700841 FOLLOWING MULTIPLE ORAL ADMINISTRATION OF MODIFIED RELEASE FORMULATION UNDER FASTED CONDITION IN PART B
Brief Title: Clinical Study to Evaluate Pharmacokinetics and Safety of PF-06700841 After Single and Multiple Oral Doses as Modified Release Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: B7931058
Record Dates: First submitted 2020-09-25; First posted 2020-10-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: Part A is a partial cross over study with 4 periods; the first three periods are IR, MR1, MR2 in fasted condition and the fourth arm is either MR1 or MR2 in fed condition.
  Part B is a multiple ascending dose study
Who Masked: Participant, Investigator
Masking Description: Part B is a sponsor open, double blind study where the investigator, medical monitor and the participants will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- PF-06700841: IR, MR1, MR2, MR1_fed (Experimental): Participants receive single doses of immediate release (IR) followed by modified release (MR) MR1 and MR2, all in fasted condition followed by MR1 in fed condition in Periods 1-4
  Interventions: Drug: PF-06700841 IR; Drug: PF-06700841 MR1; Drug: PF-06700841 MR2
- PF-06700841: MR1, MR2, IR, MR1_fed (Experimental): Participants receive single doses of MR1 followed by MR2 and IR, all in fasted condition followed by MR1 in fed condition in Periods 1-4
  Interventions: Drug: PF-06700841 IR; Drug: PF-06700841 MR1; Drug: PF-06700841 MR2
- PF-06700841: MR2, IR, MR1, MR1_fed (Experimental): Participants receive single doses of MR2 followed by IR and MR1, all in fasted condition followed by MR1 in fed condition in Periods 1-4
  Interventions: Drug: PF-06700841 IR; Drug: PF-06700841 MR1; Drug: PF-06700841 MR2
- PF-06700841: IR, MR1, MR2, MR2_fed (Experimental): Participants receive single doses of IR followed by MR1 and MR1, all in fasted condition followed by MR2 in fed condition in Periods 1-4
  Interventions: Drug: PF-06700841 IR; Drug: PF-06700841 MR1; Drug: PF-06700841 MR2
- PF-06700841: MR1, MR2, IR, MR2_fed (Experimental): Participants receive single doses of MR1 followed by MR2 and IR, all in fasted condition followed by MR2 in fed condition in Periods 1-4
  Interventions: Drug: PF-06700841 IR; Drug: PF-06700841 MR1; Drug: PF-06700841 MR2
- PF-06700841: MR2, IR, MR1, MR2_fed (Experimental): Participants receive single doses of MR2 followed by IR and MR1, all in fasted condition followed by MR2 in fed condition in Periods 1-4
  Interventions: Drug: PF-06700841 IR; Drug: PF-06700841 MR1; Drug: PF-06700841 MR2
- PF-06700841 MR3 (Dose A) or matching placebo (Experimental): Participants receive dosing regimen 1 of MR3 (Dose A) or matching placebo for 7 days under fasted condition
  Interventions: Drug: PF-06700841 MR3; Other: Placebo
- PF-06700841 MR3 (Dose B) or matching placebo (Experimental): Participants receive dosing regimen 1 of MR3 (Dose B) or matching placebo for 7 days under fasted condition
  Interventions: Drug: PF-06700841 MR3; Other: Placebo
- PF-06700841 MR3 (Dose C) or matching placebo (Experimental): Participants receive dosing regimen 1 of MR3 (Dose C) or matching placebo for 7 days under fasted condition
  Interventions: Drug: PF-06700841 MR3; Other: Placebo

INTERVENTIONS:
Drug: PF-06700841 IR — Immediate release formulation
  Arms: PF-06700841: IR, MR1, MR2, MR1_fed; PF-06700841: IR, MR1, MR2, MR2_fed; PF-06700841: MR1, MR2, IR, MR1_fed; PF-06700841: MR1, MR2, IR, MR2_fed; PF-06700841: MR2, IR, MR1, MR1_fed; PF-06700841: MR2, IR, MR1, MR2_fed
Drug: PF-06700841 MR1 — Modified release formulation 1
  Arms: PF-06700841: IR, MR1, MR2, MR1_fed; PF-06700841: IR, MR1, MR2, MR2_fed; PF-06700841: MR1, MR2, IR, MR1_fed; PF-06700841: MR1, MR2, IR, MR2_fed; PF-06700841: MR2, IR, MR1, MR1_fed; PF-06700841: MR2, IR, MR1, MR2_fed
Drug: PF-06700841 MR2 — Modified release formulation 2
  Arms: PF-06700841: IR, MR1, MR2, MR1_fed; PF-06700841: IR, MR1, MR2, MR2_fed; PF-06700841: MR1, MR2, IR, MR1_fed; PF-06700841: MR1, MR2, IR, MR2_fed; PF-06700841: MR2, IR, MR1, MR1_fed; PF-06700841: MR2, IR, MR1, MR2_fed
Drug: PF-06700841 MR3 — Modified release formulation 3
  Arms: PF-06700841 MR3 (Dose A) or matching placebo; PF-06700841 MR3 (Dose B) or matching placebo; PF-06700841 MR3 (Dose C) or matching placebo
Other: Placebo — Matching placebo
  Arms: PF-06700841 MR3 (Dose A) or matching placebo; PF-06700841 MR3 (Dose B) or matching placebo; PF-06700841 MR3 (Dose C) or matching placebo

SUMMARY:
The purpose of the study is to evaluate the pharmacokinetics (PK), safety, and tolerability of PF-06700841 following single and multiple oral doses as modified release (MR) formulations in healthy, adult participants under fasted and fed conditions. The objective of Part A is to evaluate the relative bioavailability and food effect of 2 new MR formulations, MR1 and MR2. The objective of Part B is to evaluate the PK and safety/tolerability of MR3 formulation following multiple dose administration over a 7-day period. Overall, results from both parts will facilitate further development of an MR formulation for future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants between 18 -55 years of age.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Participants who are willing and able to comply with all scheduled visits, treatment
* plan, laboratory tests, lifestyle considerations, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Conditions that affect drug absorption (e.g., gastrectomy cholecystectomy)
* History of venous and arterial thrombosis (ie, deep venous thrombosis, pulmonary embolism) or hereditary clotting disorders (in first degree immediate relatives)
* Positive urine drug test.
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of PF-06700841 in Part A | pre-dose, 1,2,4,6,8,10,12,16,24,36,48,72 hours post dose
Area under the plasma concentration-time curve from time zero to the last measured concentration (AUClast) of PF-06700841 in Part A | pre-dose, 1,2,4,6,8,10,12,16,24,36,48,72 hours post dose
Area under the plasma concentration-time curve from time zero to extrapolated infinite time (AUCinf) of PF-06700841 if data permit in Part A | pre-dose, 1,2,4,6,8,10,12,16,24,36,48,72 hours post dose
Time to reach maximum observed plasma concentration (Tmax) of PF-06700841 in Part A | pre-dose, 1,2,4,6,8,10,12,16,24,36,48,72 hours post dose
Number of participants with Treatment- Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation due to AEs in Part B | Baseline to Day 10

SECONDARY OUTCOMES:
Number of subjects with clinically relevant changes in Electrocardiogram (ECG) parameters in Part A | Pre-dose and 96 hours post dose
Number of subjects with clinically relevant changes in vital signs in Part A | Pre-dose and 96 hours post dose
Number of participants with clinically relevant changes in clinical laboratory tests in Part A | Baseline and 96 hours post dose
Number of participants with Treatment- Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Discontinuation due to AEs in Part A | Baseline to Day 4
Maximum Observed Plasma Concentration (Cmax) of PF-06700841 in Part B on Day 1 | pre-dose, 1,2,3,4,6,8,10,12,16 hours post dose on Day 1
Time to reach maximum observed plasma concentration (Tmax) of PF-06700841 in Part B on Day 1 | pre-dose, 1,2,4,6,8,10,12,16 hours post dose on Day 1
Maximum Observed Plasma Concentration (Cmax) of PF-06700841 in Part B on Day 7 | pre-dose on Day 7, 1,2,3 4,6,8,12,16,24,48,72 hours post dose on Day 7
Time to reach maximum observed plasma concentration (Tmax) of PF-06700841 in Part B on Day 7 | pre-dose on Day 7, 1,2,3 4,6,8,12,16,24,48,72 hours post dose on Day 7
Area under the plasma concentration-time curve from time zero to 24 hours (AUC24) of PF-06700841 in Part B on Day 1 | pre-dose, 1,2,4,6,8,10,12,16 hours post dose on Day 1, pre-dose on Day 3 and Day 5, pre-dose on Day 7, 1,2,3,4,6,8,12,16,24,48,72 hours post dose on Day 7
Area under the plasma concentration-time curve from time zero to 24 hours (AUCtau) of PF-06700841 in Part B on Day 7 | pre-dose, 1,2,4,6,8,10,12,16 hours post dose on Day 1, pre-dose on Day 3 and Day 5, pre-dose on Day 7, 1,2,3,4,6,8,12,16,24,48,72 hours post dose on Day 7
Terminal half-life of PF-06700841 in Part B | pre-dose, 1,2,4,6,8,10,12,16 hours post dose on Day 1, pre-dose on Day 3 and Day 5, pre-dose on Day 7, 1,2,3,4,6,8,12,16,24,48,72 hours post dose on Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Quotient Sciences, Coral Gables, Florida
  - Quotient Sciences-Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931058